CLINICAL TRIAL: NCT02916667
Title: Chrono Nutrition Intervention Program in Gestational Diabetes Mellitus
Brief Title: Chrono Nutrition (CN) Intervention Program in Gestational Diabetes Mellitus
Acronym: CN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Yoel Toledano, principal investigator, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0277-15-RMC
Record Dates: First submitted 2016-09-10; First posted 2016-09-27 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: GDM
MeSH Terms: interventions — Nutrition Policy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CNdiet (Active Comparator): CNdiet includes chrono nutritional dietary guidelines
  Interventions: Other: dietary guidelines
- GDMdiet (Placebo Comparator): GDMdiet includes regular GDM diet
  Interventions: Other: dietary guidelines

INTERVENTIONS:
Other: dietary guidelines — dietary guidelines will include chrono- nutrition diet plan

SUMMARY:
Working hypothesis and aims:

To asses Chrono Biological factors during the third trimester of gestational diabetes melittus (GDM) with birth weight and related complications. The investigators hypothesize that participants with GDM pregnancies with higher Chrono Biologocal status will be ended with higher birth weight compared to participants with GDM pregnancies with lower status. In addition, the investigators hypothesize that the Chrono Nutritional intervention program will contribute to the reduction of the rate of birth weight above percentile 90 compared with the participants with GDM in the control group.

DETAILED DESCRIPTION:
Background: Many studies have linked pre-pregnancy obesity and the metabolic syndrome, with an increased risk of developing gestational diabetes mellitus (GDM). These factors are associate with increased risk of newborn obesity, insulin resistance and diabetes. Recently, studies have shown that the "Chrono-Biological" (CB) aspects need to be considered in this context. These factors are related to endogenous circadian clocks, which regulate many body functions depending upon cycle of light and darkness during a day of almost 24 hours. By tracks daily fluctuations in heart rate, blood pressure, hormone secretion and control of a variety of metabolic pathways. Factors that can affect the setting of the circadian clock may include; Change dark and light hours, consumptions of certain nutrients during the day and more.

Chronic rhythm disruption associated with the development of obesity, diabetes, and more. Factors such as "chrono-nutrition" (CN) have a significant impact on variations in circadian rhythms includes: meals program schedule, glucose, saturated fat, caffeine and alcohol intake, and the ratio of macronutrients. Intervention studies in adults who are obese and diabetes were able to reduce the impact of these disorders by changing the composition and schedule of meals that lead to weight loss and diabetes control. Moreover, Insomnia during pregnancy can be caused by disorders CB. Insomnia affects 30-40% of all pregnancies. Some sleep disorders can be worsening by pregnancy, particularly overweight. Currently, routine monitoring and treatment of women with GDM does not include screening for sleep disorders and CN factors.

Working hypothesis and aims: To asses CB factors during the third trimester of participants with GDM pregnancies with a weight of childbirth and related complications. The investigators hypothesize that participants with GDM pregnancies with higher CB status will be ended with higher birth weight compared to participants with GDM pregnancies with a lower status.

In addition, the investigators assume that the CN intervention program will contribute to reducing the rate of birth weight above the 90 percentile compared to control group.

Methods: In a prospective cohort study, n= 280, The investigators will review the obstetric outcomes and the impact of CB disorders and complications for mother and fetus, through questionnaires. In a clinical trial n=100, The investigators will assess the effect of CN intervention on birth weight in participants with GDM pregnancies.

Expected results: Based on the investigators preliminary research and literature, The investigators expected that due to the increasing prevalence of obesity and sleep disturbance among GDM pregnancies , and the feasibility of high interference CN factors in pregnancy, Therefore, it is important to examine the impact of CB factors on maternal and fetal.

The importance of the study: Since there is a high probability that GDM is exposed to the interference of CB factors which are not monitored during GDM, this unique study, is of great importance for understanding the potential impact of the CB factors on higher birth weight rates.

ELIGIBILITY:
Inclusion Criteria:

* GDM first screened in 24-32 week of prenancy
* singleton pregnancy
* GDM screened in "Rabin medical center"
* signing an informed consent

Exclusion Criteria:

* women with history of metabolic disorder such as dislipidemia, heart disease, cancer, type 1 diabetes, type 2 diabetes, hypertension, kidney disease,liver disease, thyroids disorder, cancer.
* women with history of fertility drug therapy such as IVF or progsterone
* women who work night shifts
* women who work in air crew

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Offspring of participants with GDM with higher Chrono Biological score will be reported with higher birth weight (+100 gr) compared to offspring of participants with GDM with lower Chrono Biological score. | 2 year

SECONDARY OUTCOMES:
Offspring of participants with GDM with higher Chrono Biological score will be reported with higher birth weight above the 90 percentile compared to offspring of participants with GDM with lower Chrono Biological score. | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Moshe MI Hod, Prof, Study Director — head of the division of maternal fetal medicine at the women's hospital at Rabin medical center Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donnelly JM, Walsh JM, Byrne J, Molloy EJ, McAuliffe FM. Impact of maternal diet on neonatal anthropometry: a randomized controlled trial. Pediatr Obes. 2015 Feb;10(1):52-6. doi: 10.1111/j.2047-6310.2013.00216.x. Epub 2014 Jan 20. PMID 24443392
- [Background] Hiersch L, Yogev Y. Impact of gestational hyperglycemia on maternal and child health. Curr Opin Clin Nutr Metab Care. 2014 May;17(3):255-60. doi: 10.1097/MCO.0000000000000030. PMID 24500517
- [Background] Schellong K, Schulz S, Harder T, Plagemann A. Birth weight and long-term overweight risk: systematic review and a meta-analysis including 643,902 persons from 66 studies and 26 countries globally. PLoS One. 2012;7(10):e47776. doi: 10.1371/journal.pone.0047776. Epub 2012 Oct 17. PMID 23082214
- [Background] Yogev Y, Hiersch L. Pregnancy: impact of maternal nutrition on intrauterine fetal growth. World Rev Nutr Diet. 2014;109:101-8. doi: 10.1159/000356110. Epub 2014 Jan 16. No abstract available. PMID 24457570
- [Background] Asher G, Sassone-Corsi P. Time for food: the intimate interplay between nutrition, metabolism, and the circadian clock. Cell. 2015 Mar 26;161(1):84-92. doi: 10.1016/j.cell.2015.03.015. PMID 25815987
- [Background] Cagampang FR, Bruce KD. The role of the circadian clock system in nutrition and metabolism. Br J Nutr. 2012 Aug;108(3):381-92. doi: 10.1017/S0007114512002139. Epub 2012 Jun 8. PMID 22676899
- [Background] Tahara Y, Shibata S. Chrono-biology, chrono-pharmacology, and chrono-nutrition. J Pharmacol Sci. 2014;124(3):320-35. doi: 10.1254/jphs.13r06cr. Epub 2014 Feb 27. PMID 24572815
- [Background] Reutrakul S, Van Cauter E. Interactions between sleep, circadian function, and glucose metabolism: implications for risk and severity of diabetes. Ann N Y Acad Sci. 2014 Apr;1311:151-73. doi: 10.1111/nyas.12355. Epub 2014 Mar 14. PMID 24628249
- [Background] Jakubowicz D, Barnea M, Wainstein J, Froy O. High caloric intake at breakfast vs. dinner differentially influences weight loss of overweight and obese women. Obesity (Silver Spring). 2013 Dec;21(12):2504-12. doi: 10.1002/oby.20460. Epub 2013 Jul 2. PMID 23512957
- [Background] O'Keeffe M, St-Onge MP. Sleep duration and disorders in pregnancy: implications for glucose metabolism and pregnancy outcomes. Int J Obes (Lond). 2013 Jun;37(6):765-70. doi: 10.1038/ijo.2012.142. Epub 2012 Sep 4. PMID 22945608
- [Derived] Messika A, Toledano Y, Hadar E, Tauman R, Froy O, Shamir R. Chronobiological Factors Influencing Glycemic Control and Birth Outcomes in Gestational Diabetes Mellitus. Nutrients. 2024 Dec 31;17(1):157. doi: 10.3390/nu17010157. PMID 39796591
- [Derived] Messika A, Toledano Y, Hadar E, Shmuel E, Tauman R, Shamir R, Froy O. Relationship among chrononutrition, sleep, and glycemic control in women with gestational diabetes mellitus: a randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Sep;4(5):100660. doi: 10.1016/j.ajogmf.2022.100660. Epub 2022 May 4. PMID 35525420